CLINICAL TRIAL: NCT03658772
Title: An Open-label, Single-arm, Phase 1b Study to Evaluate the Safety and Efficacy of Grapiprant (ARY-007) in Combination With Pembolizumab in Patients With Advanced or Progressive Microsatellite Stable (MSS) Colorectal Cancer (CRC)
Brief Title: Grapiprant and Pembrolizumab in Patients With Advanced or Progressive MSS Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arrys Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARYS-001; Keynote-878 (Other: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2018-08-24; First posted 2018-09-05 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Microsatellite Stable Colorectal Cancer
Keywords: Keynote-878; ARY-007; Immuno-Oncology; checkpoint inhibitor; EP4; IK-007
MeSH Terms: interventions — grapiprant; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Cohort 1 to be enrolled before Cohort 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Single Agent run-in with grapiprant and then combination treatment of grapiprant and pembrolizumab.
  Interventions: Drug: grapiprant; Drug: grapiprant and pembrolizumab
- Cohort 2 (Experimental): Participants will be treated with grapiprant in combination with pembrolizumab.
  Interventions: Drug: grapiprant and pembrolizumab

INTERVENTIONS:
Drug: grapiprant — Cohort 1 will be treated for 1 week with oral grapiprant as a single agent, followed by 21-day combination treatment cycles of oral grapiprant in combination with IV pembrolizumab.
  Other Names: ARYS-007; IK-007
  Arms: Cohort 1
Drug: grapiprant and pembrolizumab — Cohort 2 will be administered 21-day combination treatment cycles of oral grapiprant in combination with IV pembrolizumab.
  Other Names: ARYS-007, MK3475; KEYNOTE-878; IK-007

SUMMARY:
This study will be conducted in adult participants diagnosed with any form of an advanced or progressive MSS CRC for which 1st and 2nd line standard therapy (at least one of which contained fluorouracil) is no longer effective or is intolerable. This is a phase 1b, multi-center, open label study designed to assess safety and tolerability of grapiprant in combination with pembrolizumab, to determine the recommended phase 2 dose (RP2D) with pembrolizumab, and to evaluate and characterize the PK of grapiprant alone and in combination with pembrolizumab. Disease response, pharmacodynamics, and response biomarkers will also be assessed.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female adult patients 18 years of age or older on day of signing informed consent.
* Patients must have a histologically confirmed advanced, metastatic, or progressive Microsatellite Stable (MSS) Colorectal Cancer (CRC) per institutional standards.
* Patient has received at least two prior lines of therapy for advanced or metastatic CRC, at least one of which included fluorouracil.
* Highly effective birth control.
* Measurable disease.
* Accessible tumor that can be safely accessed for multiple core biopsies and patient is willing to provide tissue from newly obtain biopsies before and during treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Adequate organ function.
* Able to swallow and absorb oral tablets.

Key Exclusion Criteria:

* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
* Current use of NSAIDs, COX-2 inhibitors and aspirin products within 3 days (preferably 7 days) before treatment initiation or at anytime during the study unless used for management of AE.
* History of severe hypersensitivity reactions to chimeric or humanized antibodies
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks prior to treatment, or 5 half-lives, whichever is shorter.
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Known active CNS metastases and/or carcinomatous meningitis.
* Active autoimmune disease that has required systemic treatment in past 2 years.
* History of non-infectious pneumonitis that required steroids or has current pneumonitis.
* Active infection requiring systemic therapy.
* Recent (within the last 12 months) or current GI ulcer, colitis or non-immune colitis.
* Known history of human immunodeficiency virus (HIV) infection, Hepatitis B, or active Hepatitis C virus infection.
* Clinically significant (i.e. active) cardiovascular disease
* Allogeneic tissue/solid organ transplant
* Medical conditions requiring concomitant administration of strong CYP3A4 or P glycoprotein inhibitors or inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of grapiprant alone and in combination with pembrolizumab | Up to 90 days after the end of treatment (average of 7 months)
  Number of incidence, severity, and duration of treatment emergent adverse events using CTCAE v5.0
Define the recommended phase 2 dose (RP2D) of grapiprant combined with pembrolizumab | Through Cycle 1 (21 days)
  Number, incidence and severity of treatment related adverse events as assessed by CTCAE 5.0

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 7 months
  Proportion of participants who achieved PR or better during the study per RECIST 1.1
Duration of Response (DOR) | 7 months
  Time when criteria for response are met, to the first documentation of relapse or progression
Progression -free survival (PFS) | Up to 12 months
  Participants who discontinue treatment without disease progression
Disease control rate (DCR) | 7 months
  Percentage of participants who achieved a CR, PR and stable disease
Overall survival (OS) | Up to 2 years from start of study drug.
  Date of study drug to date of death due to any cause. If no documentation of death at time of the analysis will be censored as of the date last known to be alive, or the data cutoff date, whichever is earlier.
Duration of treatment (DOT) | 7 months
  Time of duration on treatment
Serum tumor marker changes | 7 months
  Assess changes in serum tumor markers including but not limited to carcinoembryonic antigen (CEA), when appropriate (eg. CA-19.9, CA125, and lactate dehyrogenase (LDH)) with disease response.
Pharmacodynamic immune effects in paired tumor biopsies | predose through cycle 3 (each cycle is 21 days)
  Assess changes in tumor infiltrating helper T cells, cytotoxic T cells and regulatory monocyte/macrophages with study drug treatment
PGEM as a pharmacodynamic and predictive biomarker | PreScreening through 7 months
  Evaluate disease response in all evaluable participants and in those with a positive initial assessment of Urine prostaglandin E2 metabolite (PGEM)
PK of grapiprant: Tmax | Safety Run-in (7 days); Days 1 and 2 of first 2 cycles (every 21 days), followed by Day 1 of every even cycle beginning with cycle 4 (every 42 days) through end of treatment (average of 4 months)
  First time to reach maximum [peak] observed plasma concentration
PK of grapiprant: AUC0 last | Safety Run-in (7 days); Days 1 and 2 of first 2 cycles (every 21 days), followed by Day 1 of every even cycle beginning with cycle 4 (every 42 days) through end of treatment (average of 4 months).
  Area under the plasma concentration time curve from time 0 to the end of the dosing interval (AUC0 last)
Plasma decay half-life (t1/2) | Safety Run-in (7 days); Days 1 and 2 of first 2 cycles (every 21 days), followed by Day 1 of every even cycle beginning with cycle 4 (every 42 days) through end of treatment (average of 4 months)
  Measurement of half-life of grapiprant after dosing
Apparent oral clearance (CL/F) | Safety Run-in (7 days); Days 1 and 2 of first 2 cycles (every 21 days), followed by Day 1 of every even cycle beginning with cycle 4 (every 42 days) through end of treatment (average of 4 months)
  Rate of elimination of the drug from plasma after oral administration
Peak to trough ratio | Safety Run-in (7 days); Days 1 and 2 of first 2 cycles (every 21 days), followed by Day 1 of every even cycle beginning with cycle 4 (every 42 days) through end of treatment (average of 4 months)
  Measure how drug effect is sustained over dose interval
Observed accumulation ratio | Safety Run-in (7 days); Days 1 and 2 of first 2 cycles (every 21 days), followed by Day 1 of every even cycle beginning with cycle 4 (every 42 days) through end of treatment (average of 4 months)
  Relationship between the dosing interval and the rate of elimination for the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Santillana, MD, Study Director — Ikena Oncology; Sergio Santillana, MD, Study Chair — Ikena Oncology
Locations (4):
- United States (4):
  - Mayo Clinic Cancer Center - Scottsdale, Phoenix, Arizona
  - University of Colorado Denver-Anschutz Medical Campus, Aurora, Colorado
  - Sarah Cannon Research Institute, LLC (SCRI), Nashville, Tennessee
  - New Experimental Therapeutics of San Antonio-NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang D, Cabalag CS, Clemons NJ, DuBois RN. Cyclooxygenases and Prostaglandins in Tumor Immunology and Microenvironment of Gastrointestinal Cancer. Gastroenterology. 2021 Dec;161(6):1813-1829. doi: 10.1053/j.gastro.2021.09.059. Epub 2021 Oct 2. PMID 34606846